CLINICAL TRIAL: NCT02913378
Title: Conservative Treatment vs Locked Plate Osteosynthesis for Proximal Humerus Fractures in the Elderly: a Randomized Controlled Trial
Brief Title: Conservative vs Surgical Treatment for Proximal Humerus Fractures in the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Mauro Gracitelli, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ProxhumerusUSP
Record Dates: First submitted 2016-09-16; First posted 2016-09-23 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Shoulder Fractures
MeSH Terms: conditions — Shoulder Fractures | interventions — Fracture Fixation, Internal; Suburethral Slings

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Locking plate (Experimental): Surgical treatment with open reduction and osteosynthesis with locking plate
  Interventions: Procedure: Osteosynthesis with locking plate
- Conservative (Active Comparator): Conservative treatment with sling and rehabilitation
  Interventions: Procedure: Sling

INTERVENTIONS:
Procedure: Osteosynthesis with locking plate — Open reduction and osteosynthesis with locking plate
  Arms: Locking plate
Procedure: Sling — Conservative treatment with sling and rehabilitation
  Arms: Conservative

SUMMARY:
This is a randomized trial comparing conservative with surgical treatment (with open reduction and locking plate fixation) for proximal humeral fractures in patients aged more than 60 years.

DETAILED DESCRIPTION:
Different methods have been used in the treatment of proximal humeral fractures. Usually, treatment choice depends on fracture displacement, patient age, osteoporosis, and other characteristics. Locking plate fixation has become the most widely used method among surgical techniques, while partial arthroplasty is reserved for older patients and comminuted articular fractures. Generally, nonsurgical treatment involves a brief period with sling immobilization and physiotherapy rehabilitation.

A recent multicenter study showed no difference between conservative and surgical treatments, including internal fixation with locking plates. Two other randomized studies showed mixed results, with no relevant clinical differences between the methods. No previous trial has evaluated the quality of reduction in surgically treated fractures and its relation to outcomes. Our study aims to compare both techniques with a detailed radiographic and tomographic evaluation, in elderly patients. We also aim to evaluate the influence of reduction and plate positioning on clinical outcomes. This is a single center trial, in which surgeries will be performed by only two experienced surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Proximal humeral fractures, involving humeral head, with at least one of the following parameters:
* Head-shaft angle between 100-200° or >175° on coronal plane;
* Shaft translation (on coronal or sagittal plane) > 1cm;
* Tuberosity displacement > 0,5cm;
* Head shaft angulation >45° in axial or sagittal plane;
* Less then 30 days

Exclusion Criteria:

* No contact between shaft and humeral head
* Head-shaft angle <100° on coronal plane
* Articular head fracture with displacement > 2mm
* Fracture-dislocation
* Bilateral fracture
* Open fracture
* Ipsilateral or contralateral superior limb fracture
* Pathological fracture (tumors or bone disease, except for osteoporosis)
* Previous rotator cuff complete tear
* Previous infection
* Neurological injury
* Previous shoulder surgery
* Inability to answer subjective scores

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-07 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Individual relative Constant-Murley score | 2 years
  Constant-Murley score relative to the unaffected shoulder

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons Shoulder (ASES) score | 2 years
  Subjective functional evaluation
Constant-Murley score | 2 years
12-Item Short Form Health Survey (SF-12) | 2 years
  Quality of life evaluation
Visual analog scale (VAS) for pain | 2 years
Complication and reoperation rate | 2 years
Radiographic evaluation | 2 years
  Union, head-shaft angle, tuberosities reduction, medial support and Fjalestad reduction criteria
Rotator cuff ultrasound and magnetic resonance | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo - Department of Orthopedics and Traumatology, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196